CLINICAL TRIAL: NCT07180498
Title: The Evaluation of the Effects of Chlorhexidine and Tea Tree Oil Mouthwash on Postoperative Complications and Periodontal Healing After the Extraction of Impacted Third Molars
Brief Title: Evaluation of the Effect of Tea Tree and Chlorhexidine Mouthwashes on Healing After Third Molar Extraction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, mine alkaya karagoz, assistant professor, Harran University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HRU/25.07.49
Record Dates: First submitted 2025-09-01; First posted 2025-09-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Postoperative Complications; Trismus; Periodontal Health
Keywords: tea tree oil; third molar surgery; postoperative complications; chlorhexidine digluconate
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Trismus | interventions — chlorhexidine gluconate; Mouthwashes

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chlorhexidine group (Active Comparator): They will be instructed to gargle with chlorhexidine after brushing their teeth three times daily for 7 days.
  Interventions: Drug: Chlorhexidine Gluconate 0.12% Mouthwash
- tea tree oil group (Experimental): They will be instructed to gargle with 3 drops of tea tree oil added to 100 mL of water (approximately half a glass of water) after brushing their teeth three times daily for 7 days.
  Interventions: Drug: Tea Tree Oil mouthwash

INTERVENTIONS:
Drug: Chlorhexidine Gluconate 0.12% Mouthwash — Participants will be prescribed to gargle with chlorhexidine, which is the routine recommendation after brushing their teeth 3 times a day for 7 days after the impacted tooth extraction.
  Arms: chlorhexidine group
Drug: Tea Tree Oil mouthwash — Participants will be prescribed to gargle with tea tree oil-containing water after brushing their teeth three times a day for 7 days following the extraction of an impacted tooth.
  Arms: tea tree oil group

SUMMARY:
The purpose of this clinical study is to compare the effects of mouthwashes containing Chlorhexidine and tea tree oil on edema, pain, and trismus after the extraction of impacted third molars. Additionally, the effects on periodontal health will be examined by comparing the gum healing processes of patients using both mouthwashes.The main questions it aims to answer are:

1. Tea tree oil, said to have anti-inflammatory and antibacterial effects, could be an alternative to chlorhexidine in reducing postoperative complications after impacted tooth extraction.
2. Does tea tree oil, which has antimicrobial effects, have as positive an impact on periodontal health as chlorhexidine?Researchers will compare tea tree oil to chlorhexidine (routinely prescribed after the extraction of an impacted wisdom tooth) to see if tea tree oil works to decrease postoperative complications.

Participants will:

For 7 days after the operation, they will gargle with chlorhexidine mouthwash or mouthwash containing tea tree oil 3 times a day. They will come to the clinic for check-ups and measurements on the 2nd and 7th days after the operation. They will record their pain levels and the number of painkillers they take daily.

DETAILED DESCRIPTION:
The G x Power 3.1.9.7 program was used to calculate the sample size for this study. It was calculated that a total of 54 patients, with at least 27 patients in each group, would be included at a significance level of α=0.05 under 95% power.

Class 2 and Class B impacted third molars were selected as the ideal study group. All surgeries will be performed under local anesthesia by the same experienced oral surgeon, following standard surgical protocols. Patients will be provided with postoperative care instructions. Patients will be monitored for 7 days after surgery to assess postoperative healing. The experimental groups will receive 100% tea tree oil and a dropper. They will be instructed to gargle with 3 drops of tea tree oil added to 100 mL of water (approximately half a glass of water) after brushing their teeth three times daily for 7 days. The standard recommended antibiotic will be amoxicillin-clavulanic acid (875-125 mg, 2 tablets x 1) and paracetamol (500 mg) as a pain reliever.

The Active Comparator group will follow the standard care protocol, brushing their teeth three times daily for 7 days, followed by the use of 0.12% chlorhexidine gluconate mouthwash. The standard recommended antibiotic will be amoxicillin-clavulanic acid (875-125 mg, 2 tablets per day), and paracetamol (500 mg) will be prescribed as a painkiller.

Before the operation, measurements will be taken and recorded from the angle-labial commissure, angle-external eye angle, angle-tragus, angle-pogonion, and angle-nasal crease. The amount of plaque will be examined from all surfaces of the second molar, and the presence or absence of plaque will be noted. The patient's maximum mouth opening will be measured using a ruler. These measurements are used to compare the presence of post-operative edema and trismus.

The patient will be given a 7-day Visual Analog Scale (VAS) chart for post-extraction pain management. They will be asked to rate their pain daily for 7 days, ranging from 0 (no pain) to 10 (worst imaginable pain), and to note the number of painkillers they have used. • After tooth extraction, the patient will be called for follow-up appointments on the 2nd and 7th days. At these appointments, the patient will have plaque, maximum mouth opening, and distances between anatomical landmarks for edema assessments measured and noted.

ELIGIBILITY:
Inclusion Criteria:

* Individuals undergoing extraction of Class 2, Class B mandibular third molars impacted in the lower jaw (Pell & Gregory).
* Individuals aged 18-65.
* Individuals must be in stable general health (e.g., free of serious cardiovascular or kidney disease).
* Individuals willing to use tea tree extract or other treatments.

Exclusion Criteria:

* Individuals with a known allergy or hypersensitivity to tea tree extract.
* Individuals with serious illnesses such as heart failure or kidney disease. Patients with bleeding disorders.
* Individuals during pregnancy and breastfeeding.
* Individuals taking medications that may interact with tea tree extract (e.g., blood thinners or antihypertensives)
* Individuals previously treated for edema.
* Individuals with chronic edema.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
pain VAS measurement | preoperative, postoperative day 2, post operative day 7
  The patient will be given a chart with a 7-day VAS scale for pain control after tooth extraction. They will be asked to record their pain daily on a scale of 0 (no pain) to 10 (the worst imaginable pain) for 7 days, and to note how many painkillers they used.
amount of mouth opening | preoperative, postoperative day 2, post operative day 7
  Restriction in mouth opening for 7 days after impacted tooth extraction surgery
distance from the angulus to the labial commissure, external eye angle, tragus, pogonion, and nasal line | preoperative, postoperative day 2, post operative day 7
  The amount of facial swelling during the 7 days following impacted tooth extraction surgery

SECONDARY OUTCOMES:
Pocket depth measurement of the second molar tooth next to the extraction site and assessment of plaque presence | preoperative, postoperative day 2, post operative day 7
  The level of periodontal healing of teeth in the adjacent area during the 7 days following impacted tooth extraction surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mine alkaya karagoz, Principal Investigator — Harran University
Locations (1):
- Harran University, Faculty of Dentistry, Sanliurfa, Turkey (Türkiye)